CLINICAL TRIAL: NCT01310543
Title: RCT of the Teens and Toddlers Intervention
Brief Title: Trial of the Teens and Toddlers Intervention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TTRCT; TTRCT (Other Grant/Funding Number: Department for Education)
Record Dates: First submitted 2011-03-04; First posted 2011-03-08 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2011-04

CONDITIONS: Pregnancy in Adolescence
Keywords: Teenage pregnancy; Adolescent; Sexual health; Youth development

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teens and Toddlers (Experimental): The T&T intervention aims to prevent teenage pregnancy and promote sexual health by providing young women at risk of teenage pregnancy with regular and direct contact with a toddler and combines this with 12 modules of group-based personal-development sessions involving communication skills, anger management, discussion of positive sexual health and relationships, culminating in an accredited National Award in Interpersonal Skills. One-to-one life coaching is also provided. The intervention consists of 20 weekly afternoon sessions run in nurseries near to the secondary schools from which participating young women are recruited.
  Interventions: Behavioral: Teens and Toddlers
- Comparison (No Intervention): Girls in the comparison group will continue with their normal afternoon of schooling, which is missed by girls attending the T&T intervention for the 20 weeks of their attendance.

INTERVENTIONS:
Behavioral: Teens and Toddlers — The T&T intervention aims to prevent teenage pregnancy and promote sexual health by providing young women at risk of teenage pregnancy with regular and direct contact with a toddler and combines this with 12 modules of group-based personal-development sessions involving communication skills, anger management, discussion of positive sexual health and relationships, culminating in an accredited National Award in Interpersonal Skills. One-to-one life coaching is also provided. The intervention consists of 20 weekly afternoon sessions run in nurseries near to the secondary schools from which participating young women are recruited.
  Arms: Teens and Toddlers

SUMMARY:
Teens and Toddlers is an intervention that enables young people at risk of teenage pregnancy to spend time mentoring a toddler as well as participating in counselling and classroom work focused on youth development. This trial aims to test primary hypotheses that girls age 13/14 who are randomly allocated to participate in the T&T intervention are more likely to report use of contraception at last sex, less likely to report frequent sex without contraception over the previous 3 months, less likely to expect to become teenage parents and more likely to report high scores for youth development indicators one year after the intervention than are similar girls who are randomised not to participate. The trial involves a total of 180 girls per arm and is being conducted across England funded by the Department for Education and conducted by the London School of Hygiene and the National Centre for Social Research.

DETAILED DESCRIPTION:
1. Introduction and research questions

Although systematic reviews suggest the potential effectiveness of in-service learning (i.e. volunteering) and youth development as approaches to preventing teenage pregnancy, no intervention involving toddler-mentoring has been previously evaluated. Teens and Toddlers (T&T) is an intervention that enables young people at risk of teenage pregnancy to spend time mentoring a toddler as well as participating in counselling and classroom work focused on youth development. This trial aims to answer the following research questions:

1. What is the effect of the T&T intervention on participants' use of contraception at last sex, sex without contraception over the previous 3 months, expectation of teenage parenthood and youth development (primary outcomes) one year after intervention delivery?
2. What is the effect of the T&T intervention on participants' experience of teenage pregnancy, use of condoms at last sex, sex without condoms over the previous 3 months, emotional self-reflection and emotional vocabulary , dislike of school and knowledge of contraception (secondary outcomes) one year after intervention delivery?

2. Intervention, setting and participants

The T&T intervention is to be delivered in 22 sites in the south-east, north-east and north-west of England. Each site comprised a nursery and secondary school. Participants will be recruited in two cohorts (September 2009 and February 2010). Participants and parents will be asked to give informed consent and participating young women will be surveyed at baseline, and then randomised to intervention or control group (see below).

3. Sample size

Our power calculation focused on our primary outcome, no contraception use at last sex in the previous 6 months, which we anticipate being of 25% prevalence among our comparison group at follow-up 2, informed by the previous Ripple trial. Assuming this prevalence, in order to detect a halving of risk (in the range of effects reported by for example the Safer Choices and CAS-Carrera studies) with 80% power and 95% precision would require a sample of 180 per arm.

In addition, a further 120 girls are to be recruited at baseline to act as potential reserves should girls allocated to receive the T&T intervention drop out of the intervention in its first 8 weeks. Where such drop-out did occur, the girl dropping out of the intervention and her matched pair in the comparison group would nonetheless remain in the trial analytic sample in order to minimize selection bias. A reserve pair from the same school, one randomized to replace the drop-out on the intervention and one allocated to comparison group, would augment the drop-outs in the analytic sample. Any girls who drop out of T&T after 8 weeks will not be replaced on the intervention and will also remain in the trial analytic sample.

The sample will be recruited through the participating schools. Each school will recruit young women in groups (one or two groups per year-cohort depending on the size of the school and the level of involvement). The average size of each group will be 12 girls of whom 6 will be randomised to T&T and 6 to the control group (with an additional 4 girls recruited as reserves for every group, half of whom would if necessary be randomised to T&T and half randomised to the control group).

4. Randomisation

Within each school, girls will complete baseline assessment and be put into matched pairs based on age and sexual experience. Then they will be given a random number using a computer-based random number generator. Within each pair, the girl with the lowest number would be selected for the Teens and Toddlers programme and the girl with the highest number would be in the comparison group. The reserve pairs would be selected in a similar way, each pair would be given a random number. The two pairs with the lowest random numbers would become the reserve pairs, and the six pairs with the highest random numbers would form the main pairs for the evaluation. This randomisation process will be done using anonymised data remotely at the Offices of the National Centre for Social Research. Notification of girls' allocation will then be sent to the schools so that teachers can inform girls. Neither girls, teachers nor intervention providers can be blinded to allocation. Research data collection and analysis staff will be blinded to allocation.

5. Outcome measures

We have pre-hypothesised primary and secondary outcomes in order to avoid bias through 'data-dredging' for significant results. We have tried to balance having sufficient breadth to reflect the potentially broad benefits of participation in the T&T programme, with the need to reduce the possibility of false-positive results arising from multiple tests of statistical significance. Full questions are available on request. All measures will be piloted within an independent sample of young people who will be then interviewed regarding their understanding of the meaning of the questions and the meaning of their responses. These outcomes will be measured at follow-up 2 (72 weeks) via pen and paper self-completion questionnaire surveys done under exam conditions in a classroom supervised by two researchers with no teachers present.

6. Data collection methods

Participants will be surveyed at baseline, at the end of the programme (20 weeks) and one year after the programme is completed (72 weeks). Girls will be offered £10 vouchers to girls in intervention and comparison group for completion of questionnaires. A repeat visit to schools will be made to survey those students missing the previous visit. Multiple forms of contact information will also be taken so that students repeatedly missing from, or moving, school can be tracked down.

7. Analysis

There is no plan for an interim analysis done to inform whether stopping rules should be implemented because by the time an analysis of follow-up 2 data for cohort 1 is available then cohort 2 will already have experienced the intervention. Analysis of effects estimates will be done on an 'intention to treat' basis with all participants and controls originally recruited to the study plus any reserves brought into the programme to augment drop-outs being included in the analysis regardless of attendance in the programme. Logistic regression will be used to estimate effect sizes for binary outcomes and ANOVA for continuous measures. Each will generate crude and adjusted estimates, the latter adjusting for any significant (P<0.1) baseline differences in socio-demographic measures or baseline values of outcome measures.

8. Governance

The trial will be managed by an executive group consisting of researchers from the National Centre for Social Research and the London School of Hygiene and Tropical Medicine which will meet monthly. The Trial Steering Group function will be fulfilled by a committee comprising representatives from each research team, the funders (Department for Education), the providers (Teens and Toddlers) as well as two independent members (Meg Wiggins, Senior Research Fellow, Social Science Research unit, Institute of Education and Sally Hopewell, Senior Research Fellow, Centre for Statistics in Medicine, University of Oxford). This group will meet quarterly to scrutinise trial design and methods and assess data quality. This group will thus including within its function that of a data monitoring committee.

ELIGIBILITY:
Inclusion Criteria:

1. Young women age 13/14
2. Perceived by teachers as:disengaged from or uninterested in school; not working to their potential in school; exhibiting poor or disruptive behaviour in class; having a poor attendance record; parents rarely/never attending parents' evenings; parent or sibling being a teenage parent; and/or being currently/previously in care

Ages: 13 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 449 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Use of contraception at last sex | 72 weeks
  Self-report measure based on pen and paper questionnaire

SECONDARY OUTCOMES:
Frequency of sex without contraception over the previous 3 months | 72 weeks
  Also self-report (N.B. Because of the broad aims of the intervention this outcome is being treated as a primary outcome also)
Expectation of teenage parenthood | 72 weeks
  Also self report (N.B. Because of the broad aims of the intervention this outcome is being treated as a primary outcome also)
Youth development | 72 weeks
  Composite score derived from scaled items (N.B. Because of the broad aims of the intervention this outcome is being treated as a primary outcome also)
Teenage pregnancy | 72 weeks
  Self-report
Use of condoms at last sex | 72 weeks
  Self-report
Sex without condoms over the previous 3 months | 72 weeks
  Examines episodes of sex without condom use via self report measure
emotional self-reflection | 72 weeks
  Self report
Emotional vocabulary | 72 weeks
  Self-report
Dislike of school | 72 weeks
  Self report
Knowledge of contraception | 72 weeks
  Composite score drawing on several self-report items
Doesn't positively like self | 72 weeks
  Self-report
Believes best age to have sex <16 | 72 weeks
  Self report
Attitude to unprotected sex | 72 weeks
  Self report
Believes it would be difficult to talk openly about sex with boyfriend | 72 weeks
  Self report
Believes it would be difficult to talk about the pill in clinic or with doctor | 72 weeks
  Self report

CONTACTS AND LOCATIONS:
Overall Officials: Chris Bonell, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- National Centre for Social Research, London, London, United Kingdom